CLINICAL TRIAL: NCT05432544
Title: A Phase 1, Randomized, Double Blind, Dose-escalation, Placebo Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Subcutaneous Injection of SHR-1918 Injection in Healthy Subjects
Brief Title: Safety and Tolerability of SHR-1918 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SHR-1918-101
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Hyperlipemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: SHR-1918 injection compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAD, SHR-1918 (Experimental): Up to 6 cohorts of healthy subjects will receive a single dose of SHR-1918 injection
  Interventions: Drug: SHR-1918
- SAD, SHR-1918 placebo (Placebo Comparator): Up to 6 cohorts of healthy subjects will receive a single dose of SHR-1918 placebo injection
  Interventions: Drug: SHR-1918 placebo

INTERVENTIONS:
Drug: SHR-1918 — Ascending dose
  Arms: SAD, SHR-1918
Drug: SHR-1918 placebo — Ascending dose
  Arms: SAD, SHR-1918 placebo

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of SHR-1918 injection in healthy subjects. In addition, this study will provide information on pharmacokinetics and pharmacodynamics of SHR-1918 injection in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤65 on the date of signing the informed consent, males or females;
2. 1.7 mmol/L≤TG≤5.6 mmol/L，2.6 mmol/L≤LDL-C<4.9 mmol/L;
3. Understand the study procedures and methods, volunteer to participate in the study, and sign the informed consent.

Exclusion Criteria:

-

1.History of disease or treatment for:

1. Known allergic reaction to experimental drugs or severe allergic reaction to other antibody drugs;
2. Malignncy;
3. Combined cardiovascular, hepatic, renal, gastrointestinal, neuropsychiatric, hematological, or metabolic diseases;
4. History of any drug use prior to screening or within 2 weeks prior to baseline

2.Any one of the following tests at screening :

1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or gamma-glutamyl transferase (GGT) exceeding 2 times ULN, or total bilirubin exceeding 1.5 times ULN
2. Creatine kinase (CK) exceeding 3 times the upper limit of normal (ULN)

3.General:

1. History of drug or substance abuse;
2. Average of 5 or more cigarettes per day during the 4 weeks prior to screening;
3. History of blood donation within 3 months prior to screening, or severe blood loss (≥400 mL blood loss), or received a blood transfusion within 4 weeks;
4. Vaccination within 2 weeks prior to screening or planned during the course of the trial

4.The Investigator determines that the subjects have poor compliance or have any factors that may prevent them from participating in the study, including, but not limited to, the study placing the subjects at unacceptable risk or possibly interfering with the study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-12-11 (Estimated); Study Completion 2023-12-12 (Estimated)

PRIMARY OUTCOMES:
To assess the number of subjects with adverse events (AEs) | up to day 190
To assess the number of subjects with serious adverse events (SAEs) | up to day 190

SECONDARY OUTCOMES:
To assess AUC0-t | up to day 190
To assess AUC0-∞ | up to day 190
To assess Tmax | up to day 190
To assess Cmax | up to day 190
To assess t1/2 | up to day 190
To assess CL/F | up to day 190
To assess 、V/F. | up to day 190
To assess LDL-C | up to day 190
To assess TC | up to day 190
To assess HDL-C | up to day 190
To assess TG | up to day 190
To assess ApoB | up to day 190
To assess ApoA1 | up to day 190
To assess Lp(a) | up to day 190
To assess VLDL-C. | up to day 190
To assess ADA(or/and Nab). | up to day 190

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Qin R, Ye L, Duan L, Li M, He W, Mei X, Li D, Jin R, Lv C, Zhu M, Wang S, Xie Z. SHR-1918, A Monoclonal Antibody Against Angiopoietin-Like 3, in Healthy Subjects: A Randomized, Double-Blind, Placebo-Controlled Study. Clin Pharmacokinet. 2025 Aug;64(8):1245-1253. doi: 10.1007/s40262-025-01539-8. Epub 2025 Jun 27. PMID 40576753